CLINICAL TRIAL: NCT04586608
Title: Administration of an Intravenous Fat Emulsion Enriched With MCT/ω-3 Fatty Acids is Beneficial Towards Anti-inflammatory Related Fatty Acid Profile in Preterm Neonates: a Randomized, Double-blind Clinical Trial.
Brief Title: Investigation of Administration of MCT/ω-3 Fatty Acids is Towards Anti-inflammatory Related Fatty Acid Profile in Preterm Neonates.
Acronym: MCT/ω-3 FA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iaso Maternity Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, Panos Papandreou, pharmD PhDc Head of Parenteral Nutrition Unit, Iaso Maternity Hospital, Athens, Greece
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201802
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active comparator (Active Comparator)
  Interventions: Dietary Supplement: MCT/ω-3 fatty acids
- soybean oil-based IVFE (Other): soybean oil-based IVFE
  Interventions: Dietary Supplement: soybean oil-based IVFE

INTERVENTIONS:
Dietary Supplement: MCT/ω-3 fatty acids — The provision of ω-3 fatty acids to premature neonates in the Parenteral Nutrition.
  Arms: active comparator
Dietary Supplement: soybean oil-based IVFE — soybean oil-based IVFE
  Arms: soybean oil-based IVFE

SUMMARY:
Intravenous administration of pure soybean oil emulsions high in linoleic acid may lead to inflammation and lipid peroxidation in preterm neonates. The aim of the present study was to investigate the effects of a medium-chain triglyceride (MCT)/n-3 polyunsaturated fatty acid (PUFA)-enriched intravenous fat emulsion (IVFE) on plasma fatty acid (FA) profile in preterm neonates. Methods: In this double-blind randomized study, 92 preterm neonates (gestational age <32 weeks, birth weight <1500g) were assigned to receive either MCT/n-3 PUFA-enriched IVFE (Intervention Group) or soybean oil-based IVFE (Control Group). Neonates' parents gave their informed written consent for inclusion in the study. Levels of FAs were measured at baseline (day 0) and day 15 of parenteral nutrition with gas-chromatography mass-spectrometry.

ELIGIBILITY:
Inclusion Criteria:

Preterm neonates with gestational age <32 weeks

* birth weight <1500 g
* admitted to a tertiary neonatal intensive care unit within 12 hours after birth

Exclusion Criteria:

* anticipated needs for parenteral nutrition (PN) at ˃70% of total daily energy for <10 days evidence of intrauterine infection,
* perinatal asphyxia
* major congenital anomalies
* refusal of parental consent

Ages: 0 Days to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Alterations on Metabolic Fatty Acid Profile of the Premature Neonates | two years
  the detection of clinically significant differences in plasma n-3 PUFAs, n-6 PUFAs and EPA in the MCT/ω-3 PUFA-enriched IVFE group compared to the SO-IVFE group post intervention.
  the detection of clinically significant differences in plasma n-3 PUFAs, n-6 PUFAs and EPA in the MCT/ω-3 PUFA-enriched IVFE group compared to the SO-IVFE group post intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Panos Papandreou, Athens, Greece